CLINICAL TRIAL: NCT01882582
Title: Evaluation of Immune Signaling Networks in Healthy Human Volunteers
Status: Completed | Type: Observational
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 25292
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Normal Immune Cell Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand whether and to what extent the activity of immune cells in blood varies over time under normal conditions as assessed in healthy subjects. Results of this study will provide the foundation for helping us evaluate changes in immune cell activities in response to surgery and drugs used in anesthesia. The overall purpose of our research is to understand immune health in the context of anesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Good general health

Exclusion Criteria:

1. Recent cold or flu
2. Chronic use of medications affecting the immune system
3. Chronic illness
4. Smoking habit
5. History of drug abuse
6. Current recreational drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population consists of a community sample.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Numerical and functional changes of circulating immune cells over time in healthy individuals | Day 1, Day 2, Day 7, Day 28
  This is an exploratory study. Numerical and functional (phosphorylation of signaling molecules and transcription factors) behavior of all circulating immune cells will be captured. Blood specimens collected at referenced time points will be analyzed with mass cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University SOM
Locations (1):
- Stanford University, Stanford, California, United States